CLINICAL TRIAL: NCT04777162
Title: Efficacy and Safety of Tislelizumab Plus Anlotinib in PD-1/PD-L1 Resistant Metastatic Gastric or Colorectal Cancer: a Single Arm Phase II Clinical Trial
Brief Title: Tislelizumab Plus Anlotinib for Immunotherapy Resistant Gastrointestinal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Professor, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tislelizumab plus Anlotinib
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Gastric Cancer; Colo-rectal Cancer
MeSH Terms: conditions — Stomach Neoplasms; Colonic Neoplasms | interventions — tislelizumab; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tislelizumab+anlotinib (Experimental): patients will be administrate with dual drugs, tislelizumab plus anlotinib.
  Interventions: Drug: Tislelizumab; Drug: Anlotinib

INTERVENTIONS:
Drug: Tislelizumab — For included participants, tislelizumab would be administrated 200mg q3w iv.
Drug: Anlotinib — Patients will be administrated with Anlotinib 12mg p.o. d1-d14 q3w.

SUMMARY:
Immunotherapy acquired resistance was observed in clinical practice. The investigators intended to add anlotinib to PD-1 inhibitors, hoping reverse the resistance.

DETAILED DESCRIPTION:
Anti-angiogenesis seems have positive effects on tumor immune microenvironment. the combination of PD-1/PD-L1 inhibitors and TKIs exhibited favorable efficacy on gastrointestinal malignancies. Here the investigators want to examine the efficacy and survival benefit from the combination therapy to PD-1 acquired resistance patients, which turns out to be critical issues in recent years.

ELIGIBILITY:
Inclusion Criteria:

* ECOG scored 0 or 1, ≥18 years old, expected OS≥3 months;
* Histology confirmed unresectable or metastatic gastric/gastroesophageal junction adenocarcinoma or colorectal cancer;
* ≥1 evaluable lesion based on RECIST 1.1;
* Patients received PD-1/PD-L1 in the last treatment line, and should meet following conditions:

  i) there was no severe immune-related adverse events, ii) the duration between tumor progression and screening should be 3-12 weeks, iii) the best evaluation results should be PR or CR when receiving PD-1/PD-L1 treatment but progression was confirmed in the latest evaluation, iv) patients were diagnosed with special pathology subtypes, that are sensitive to immunotherapy, such as dMMR, MSI-H tumors, or gastric cancer with PD-L1 CPS≥10, PFS≥6 months in the last treatment line;
* laboratory test should meet following standard: i) HB≥90g/l, neutrophils≥1.5*10^9/L, plt≥100*10^9, ii) ALT and AST<2.5xULN (5ULN for liver metastatic patients), TBIL≤2×ULN, Cr≤1.5×ULN, and Ccr>50μmol/L iii) APTT, INR and PT≤1.5×ULN iv) LVEF≥50%
* for female participants, Hcg should be negative and both male and female participants should have contraception measures
* participants should be informed consent, and voluntary.

Exclusion Criteria:

* received anlotinib or other TKIs previously;
* allergic to other monoclonal antibody before the treatment;
* diagnosed with other malignancy in last five years (cured skin basal carcinoma, prostate cancer or cervical caner in situ were excluded)
* concurrent with other active autoimmune disease;
* any condition that require immune suppressor, such as cortisol (>10mg/d prednisone equally), CTX;
* conditions affect oral absorption (eg: dysphagia, intestinal obstruction; chronic diarrhea);
* uncontrolled pleural effusion, hydropericardium and seroperitoneum;
* brain metastasis;
* received other anti-tumor treatment in past 3 weeks, eg: surgery, radiotherapy, target therapy, immunotherapy, and traditional Chinese therapy (target therapy less than 5 half-life period, 5-Fu less than 14 days were excluded);
* concurrent with uncontrolled other diseases, i) hypertension (>150/90mmHg) ii) unstable angina pectoris, ≥ level 2 heart failure, arrhythmia within last 6 months; iii) clinical meaningful liver disease, eg: active HBV/HCV hepatitis; iv) HIV positive; v) uncontrolled diabetes; vi) urine protein ≥++ or 24h urine protein >1g;
* injected vaccine in past 4 weeks, or administrated with antibiotics;
* investigator assumed improper conditions, such as mental disease, family or society factors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 2 years
  the rate of patients reached PR or CR based on RECIST 1.1

SECONDARY OUTCOMES:
progression-free survival | Up to 2 years
  the time from recruiting to death or progression
overall survival | Up to 2 years
  the time from recruiting to death

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No